CLINICAL TRIAL: NCT03637296
Title: Adapting Critical Time Intervention to Support Inpatient Medical Care Transition
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is terminated due to COVID-19 pandemic
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Healthfirst (Other); Montefiore Medical Center (Other); Bronx-Lebanon Hospital Center Health Care System (Other)
Responsible Party: Principal Investigator, Tom Smith, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7657
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Medical Complication
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Prospective cohort with comparison group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Critical time intervention (Experimental): Individuals who receive intensive care management during and following discharge from the inpatient medical unit.
  Interventions: Other: Critical time intervention
- Treatment as usual (No Intervention): Individuals who receive routine care management during and following discharge from the inpatient medical unit.

INTERVENTIONS:
Other: Critical time intervention — Care management offered by individual with experience working with individuals with serious mental illness. The care managers engage individuals before they are discharged from the hospital and work with them in the community to support linkages with medical and behavioral health care providers. Care managers provide problem-solving, advice, and support to maximize patients' engagement in care.
  Arms: Critical time intervention

SUMMARY:
We are pursuing a pilot study to assess the feasibility and preliminary effectiveness of adapting a critical time intervention (CTI) approach for adults with schizophrenia who have been admitted for the inpatient treatment of ambulatory care sensitive conditions. These are common health conditions, such as chronic obstructive pulmonary disease or short-term complications from diabetes mellitus, in which appropriate ambulatory care prevents or reduces the need for inpatient treatment. A 2-arm pilot study will randomize 80 eligible inpatients to receive either: 1) treatment as usual (TAU) (N=20); or 2) CTI and TAU (N=40). Participants assigned to CTI will meet with a CTI care manger during their inpatient stay and over a 3-month period following hospital discharge. CTI care managers will assess and address patient needs and barriers to outpatient medical and mental health care and provide support and assistance with health and mental health care management. The primary outcome measure will be all-cause hospital readmissions at 7 and 30 days following discharge. Secondary outcomes will include follow-up with medical and mental health at 7 and 30 days following hospital discharge. Patients receiving CTI will also receive 6 and 12 week assessments to evaluate secondary outcomes including satisfaction with CTI services, psychiatric symptoms, community function, and involvement in medical care decisions.

DETAILED DESCRIPTION:
For adults with schizophrenia, the transition from hospital inpatient to outpatient care poses substantial risks of treatment disengagement. Traditional case management approaches for patients with schizophrenia have involved telephonic follow-up after discharge from inpatient mental health care and have yielded poor results. Much less information exists regarding outcomes for patients with schizophrenia discharged following inpatient medical care. Given that these patients often have difficulty accessing and adhering to medical treatments, patients with schizophrenia who are admitted to a hospital for treatment of a medical condition are especially vulnerable to failed care transitions. Intensive interventions involving home visits, social support, motivational interviewing, and accompanying patients to outpatient appointments have shown positive results for patients discharged following inpatient mental health care, and may therefore be effective for patients with schizophrenia discharged following inpatient medical care. Critical Time Intervention (CTI) is a novel evidence based time-limited intervention that involves ongoing community-based contacts with patients from trained care managers to facilitate connections to aftercare providers and community and support systems following hospital discharge. This pilot study will adapt CTI for use with patients with schizophrenia who are admitted to one of 2 safety net hospitals in Bronx, New York, for treatment of ambulatory care sensitive conditions (medical conditions for which appropriate ambulatory care should limit the need for inpatient treatment). We will randomize 80 eligible inpatients to receive either: 1) treatment as usual (TAU) (n=20); or 2) CTI and TAU (n=40). During a 3-month period prior to randomization, an Adaptation Team of research and hospital staff will review data from qualitative interviews of clinical staff and patients to identify factors likely to facilitate and impede CTI implementation. The team will then adapt the CTI to increase the likelihood of successful implementation. In the randomization phase, participants assigned to CTI will meet with a CTI care manger during their inpatient stay and over a 3-month period following hospital discharge. CTI care managers will assess and address patient needs and barriers to outpatient medical and mental health care and provide support and assistance with medical and mental health care management. For quantitative analyses, the primary outcome measures will be all-cause hospital readmissions at 7 and 30 days following discharge. Secondary outcomes will include follow-up with medical and mental health outpatient care at 7 and 30 days following hospital discharge. Patients receiving CTI will also be assessed to evaluate satisfaction with CTI services, psychiatric symptoms, community function, and involvement in medical care decisions. The proposed study will test whether a time-limited novel intervention helps overcome common barriers to adherence with outpatient medical and mental health care and reduces hospital readmissions for a vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 64 years old
* Diagnosis of schizophrenia
* Admitted to medical unit at collaborating hospital
* Admission diagnosis of Ambulatory Care Sensitive Condition

Exclusion Criteria:

* Not enrolled in Healthfirst Medicaid Managed Care plan for 12 months prior to admission

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Smith, MD, Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - Bronx Care Health System, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be made available for research to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with public repositories including the National Database for Clinical Trials related to Mental Illness (NDCT). Data will include baseline demographic data, and baseline and post raw data derived from functioning and symptom measures.
Supporting Information: Study Protocol
Time Frame: A list of all data expected to be collected in the project will be submitted within 6 months of award. Subsequently, descriptive and raw data will be submitted on a semi-annual basis. Unpublished de-identified data will be submitted prior to study completion and will be shared within one year after project completion, or when the data are published, whichever is earlier.
Access Criteria: Data in NIH repositories may be accessed through the NIH Data Access Committee which reviews data access and submission requests.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Critical Time Intervention | Treatment as Usual
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Critical Time Intervention | Treatment as Usual | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (9.4) | 45.5 (5.8) | 49.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: 7 Days Hospital Inpatient All-cause Readmission Rates
Description: Rates of hospital inpatient readmission within 7 days following discharge
Time Frame: Within 7 days following discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Critical Time Intervention | Treatment as Usual
Number analyzed (Participants) | 10 | 5
Participants | 3 | 0

2. Primary Outcome: 30 Days Hospital Inpatient All-cause Readmission Rates
Description: Rates of hospital inpatient readmission within 30 days following discharge
Time Frame: Within 30 days following discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Critical Time Intervention | Treatment as Usual
Number analyzed (Participants) | 10 | 5
Participants | 7 | 0

3. Secondary Outcome: Number of Participants Who Follow up With Outpatient Medical Within 7 Days of Hospital Discharge
Description: Number of Participants who follow-up with outpatient medical attendance within 7 days of hospital discharge at follow-up appointments
Time Frame: Within 7 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Critical Time Intervention | Treatment as Usual
Number analyzed (Participants) | 10 | 5
Participants | 7 | 4

4. Secondary Outcome: Number of Participants Who Follow-up With Outpatient Medical Within 30 Days of Hospital Discharge
Description: Number of Participants who follow-up with outpatient medical attendance within 30 days of hospital discharge at follow-up appointments
Time Frame: Within 30 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Critical Time Intervention | Treatment as Usual
Number analyzed (Participants) | 10 | 5
Participants | 9 | 4

5. Secondary Outcome: Number of Participants Who Follow-up With Outpatient Mental Health Services Within 7 Days of Hospital Discharge
Description: Number of Participants who follow-up with Outpatient Mental Health Services attendance within 7 days of hospital discharge at follow-up appointments
Time Frame: Within 7 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Critical Time Intervention | Treatment as Usual
Number analyzed (Participants) | 10 | 5
Participants | 1 | 0

6. Secondary Outcome: Number of Participants Who Follow-up With Outpatient Mental Health Services Within 30 Days of Hospital Discharge
Description: Number of Participants who follow-up with Outpatient Mental Health Services attendance within 30 days of hospital discharge at follow-up appointments
Time Frame: Within 30 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Critical Time Intervention | Treatment as Usual
Number analyzed (Participants) | 10 | 5
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Critical Time Intervention | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03637296/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT03637296/SAP_001.pdf
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03637296/ICF_002.pdf